CLINICAL TRIAL: NCT03565510
Title: A Randomized, Controlled, Cross-over Trial Investigating the Impact of a High-protein Diet on Energy Metabolism in Healthy Men
Brief Title: The Impact of a High-protein Diet on Energy Metabolism in Healthy Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Almased Wellness GmbH (Industry)
Responsible Party: Principal Investigator, Carla Prado, Assistant Professor / CAIP Chair in Nutrition, Food and Health, CIHR New Investigator, University of Alberta
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00083005
Record Dates: First submitted 2018-06-11; First posted 2018-06-21 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Dietary Modification
Keywords: High-protein diet; Energy metabolism
MeSH Terms: interventions — Diet, High-Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Those assigned to the Control group will receive a diet composed of 55% of carbohydrate, 15% of protein, and 30% of lipid (similar to the North American dietary pattern).
- High-Protein Diet (Experimental): Those assigned to the High-Protein Diet group will receive a diet composed of 35% of carbohydrate, 40% of protein, and 25% of lipid constructed around a soy protein-based total diet replacement.
  Interventions: Dietary Supplement: High-Protein Diet

INTERVENTIONS:
Dietary Supplement: High-Protein Diet — The high-protein diet is composed of 35% of carbohydrate, 40% of protein, and 25% of lipid constructed around a soy protein-based meal replacement.
  Arms: High-Protein Diet

SUMMARY:
The aim of this study is to investigate the impact of a high-protein diet (achieved with the use of a nutritional supplement, Almased®) versus a diet of a typical North American macronutrient distribution on energy metabolism, metabolic blood markers and appetite sensations.

This study will be a randomized, controlled, cross-over trial of an acute nutritional intervention. A total of 20 participants will be randomly assigned (1:1) to one of the following groups:

* Control group (CON).
* High protein diet group (HP).

The diets given to participants in both groups will be eucaloric.

While receiving the diets in the whole body calorimetry unit for 32 hours, participants' overall changes in energy metabolism, metabolic blood markers, and appetite sensations will be assessed.

DETAILED DESCRIPTION:
This study will be a randomized, controlled, cross-over trial of an acute nutritional intervention. The participants will be randomly assigned (1:1) to one of the following groups:

* Control group (CON). Those assigned to the CON will receive a diet composed of 55% of carbohydrate, 15% of protein, and 30% of lipid (similar to the North American dietary pattern [3]).
* High protein diet group (HP). Those assigned to the HP will receive a diet composed of 35% of carbohydrate, 40% of protein, and 25% of lipid constructed around a soy protein-based meal replacement (Almased®).

The diets given to participants in both groups will be eucaloric.

The following metabolic changes will be assessed between the diets:

* Energy metabolism (energy expenditure and substrate oxidation);
* Metabolic blood markers [glucose, insulin, lipid panel, peptide tyrosine-tyrosine (PYY), glucagon-like peptide-1 (GLP-1), ghrelin, leptin, free glycerol, and free fatty acids];
* Appetite sensations (hunger, satiety, fullness, and prospective food consumption).

Sample Size: A total of 18 participants will be able to detect an effect size of 1.41. The effect size was calculated based on changes in RQ (0.90 ± 0.04 in control group and 0.85 ± 0.03 in a high protein group) from a previously published study. Accounting for a 20% attrition rate (formula N=18/1-20%), the total sample size of 23 participants will have a power of 80% with a significance level of 5%. The sample size calculation was done using G*Power version 3.1.9.2.

Visit # 1 - Screening Visit: During the screening visit, the study coordinator will run through the study protocol and obtain written informed consent as well as participants' contact information. Eligibility to participate in the study will be based on set inclusion and exclusion criteria, completion of physical activity questionnaires, anthropometric assessment, bioelectrical impedance analysis (BIA), and analysis of biomarkers for kidney and liver function, electrolyte status, and thyroid-stimulating hormone.

Visit # 2 - Orientation Visit: During the orientation visit, participants will answer questions related to their health status and food preferences, will have their energy requirements assessed by an 1-hour WBCU test and will be provided an explanation about the run-in diet period. Body composition will also be assessed using dual energy X-ray absorptiometry (DXA) and air displacement plethysmography (ADP).

Visits # 3 & 5 - Fitness Test & Run-In Diet Visit: To standardize the exercise intensity while in the WBCU, participants will attend a fitness test visit prior to their first WBCU test visit. They will perform a submaximal exercise test on a treadmill (Freemotion Incline Trainer). The exercise test will begin at an individualized walking speed characterized as comfortable and sustainable. The incline will increase by 2% every three minutes until a RER of 0.9 has been achieved. During exercise, expired gases will be analyzed by a calibrated TrueMax® metabolic measurement system (ParvoMedics, Sandy, UT). To reproduce the same conditions during the WBCU exercise session, a breakfast identical to that provided inside the WBCU (CON Group) will be given to participants at 9 am and the treadmill test will start at 10:20 am. To determine the workload for the WBCU exercise session, each participant's respiratory exchange ratio (RER) will be plotted against their fitness test workload. The workload at which an RER of 0.85 occurred will be selected as the workload for the WBCU. We anticipate there will be a RER of 0.85 ± 0.03 during the WBCU control exercise session. The small difference may be due to factors such as the change in substrate oxidation throughout a 40-minute bout of exercise.

After the fitness test, participants will receive all the meals necessary to complete the 3-day run-in diet. This will standardize dietary intake among participants and minimize the effects of any eating style/behaviours on baseline data. The run-in diet will be a eucaloric diet and will have the same macronutrient distribution as of CON group diet (55% of carbohydrate, 15% of protein, and 30% of lipid). During this three-day run-in diet period, participants will be asked to abstain from any strenuous exercise, including endurance and/or resistance exercises. They can exercise (moderate) and drink coffee during the first and second days of run-in diet, but not during the third day.

Visits # 4 & 6 - Whole Body Calorimetry Test Visits: Participants will complete a WBCU test visit twice during the study period, which will occur after the run-in diet periods. These visits will consist of two 32 hours (1.5 days) energy expenditure assessments inside the WBCU. During the 32-hour measurement period, participants of both groups (CON and HP) will be provided with a five-meal diet (breakfast, lunch, dinner, and two snacks) through an air-lock drawer system. The CON group will receive a diet composed of 55% of carbohydrate, 15% of protein, and 30% of lipid. The participants will receive breakfast, lunch, dinner and two snacks (afternoon and evening). The HP group will receive a diet composed of 35% of carbohydrate, 40% of protein, and 25% of lipid constructed around a soy protein-based meal replacement (Almased®). Participants will consume approximately 1 gram of Almased® per kg of body weight mixed with olive oil and low-fat milk (1% fat) in their breakfast, lunch and dinner. Two snacks (afternoon and evening) composed of approximately 1 gram of Almased® per kg of body weight mixed with apple juice and olive oil will also be provided. Amounts of low-fat milk, olive oil, and apple juice will be adjusted on an individual basis in order to achieve the desired macronutrient composition for the HP group. A variation of ± 2% for each macronutrient and ± 50 kcal/day will be considered.

The exercise session will be performed on the first morning (from 10:20 a.m. to 11:00 a.m.) spent in the WBCU. The session will be performed on a treadmill (BH T10 Pro Treadmill). The speed and grade of the treadmill will be set based on the fitness test as previously described.

Blood samples will be taken four times while participants are in the WBCU:

* Fasting on the first day (at 07:45 a.m.);
* After the exercise session on the first day (at 11:00 a.m.);
* Two hours postprandial on the first day (at 02:30 p.m.);
* Fasting on the second day (at 08:30 a.m.). The following blood markers will be analysed: glucose, insulin, lipid panel, PYY, GLP-1, ghrelin, leptin, free glycerol, and free-fatty acid. While participants are inside the WBCU, urine must be collected during the entire time. This is necessary to determine total nitrogen excretion, protein used by participant's body during the test day. Participants will be asked to rate their appetite sensations on a 100-mm visual analogue scale (VAS) immediately before and 30 minutes after each meal and snack provided in the WBCU in order to measure subjective appetite sensations (hunger, satiety, fullness, and prospective food consumption). Participants will be asked to wear an accelerometer around the wrist during sleep. The motion sensor will measure participants' activity patterns during sleep. A two week wash-out period between the WBCU test visits is needed to reduce the carryover effects of the interventions. A two week washout period is typical of feeding trials with soy isoflavone intervention [4, 5].

Statistical Analyses: Data distributions will be evaluated by the Shapiro-Wilk W-test. Parametric variables will be expressed in average and standard deviation and then converted into delta scores (i.e. post-pre values). To determine the differences among the variables analyzed after the intervention (within) and between CON and HP groups (between), Student's t-test or Mann-Whitney tests will be applied, according to data distribution. Pearson's correlation coefficients will be determined to assess whether there is a statistically significant correlation among the variables. All analyses will be performed using SPSS version 22.0, considering a critical significance value of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Healthy;
* Non-smoker;
* Male;
* Aged 18 to 34.9 years;
* BMI between 18.5 and 24.9 kg/m² (preferably between 20 and 24.9 kg/m2);

Exclusion Criteria:

* Have previously been diagnosed with any chronic disease;
* Are taking any medications which may alter energy metabolism or body composition (exception: if taking antidepressants in a stable dose for > two months);
* Are lactose, gluten and/or soy allergic/intolerant;
* Follow a vegetarian, vegan or restrictive dietary pattern;
* Have used nutritional supplements in the past two months (except micronutrients);
* Are performing or have performed over an hour per day of leisure time physical activity or more than seven hours per week of strenuous activity in the past three months;
* Have had a nuclear medicine scan or injection of an X-ray dye in the past week;
* Have had a barium test/exam in the last two weeks;
* Suffer from claustrophobia.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Difference in fat balance assessed by indirect calorimetry during 32 hours of a high-protein (HP) total diet replacement compared to 32hours of a control (CON) diet. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  To measure the differences in fat balance during 32 hours of a high-protein (HP) total diet replacement compared to 32hours of a control (CON) diet.

SECONDARY OUTCOMES:
Difference in 24-hour energy expenditure assessed by indirect calorimetry during 32 hours of a high-protein (HP) total diet replacement compared to 32hours of a control (CON) diet. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  To measure the differences in 24-hour energy expenditure during 32 hours of a high-protein (HP) total diet replacement compared to 32 hours of a control (CON) diet.

OTHER OUTCOMES:
Changes in appetite sensations assessed by a 100 mm visual analogue scale questionnaire. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  Changes in hunger, satiety, fullness, and prospective food consumption will be rated by participants on a 100 mm visual analogue scale immediately before and 30 minutes after each meal and snack provided while participants spend 32 hours inside the whole body calorimetry unit while receiving a high-protein diet or a control diet. The 100 mm visual analogue scale is administered using the paper-and-pen method and participants are instructed to make a single vertical mark at the appropriate point between the two anchors on each scale to indicate the intensity of their subjective states regarding each element (between 0 and 100 mm):
  Hunger: 0 mm = "I am not hungry at all"; 100 mm = "I have never been more hungry".
  Satiety: 0 mm = "I am completely empty"; 100 mm = "I cannot eat another bite". Fullness: 0 mm = "Not at all full"; 100 mm = "Totally full". Prospective food consumption: 0 mm = "Nothing at all"; 100 mm = "A lot".
Changes in blood glucose levels. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  Changes in glucose will be assessed four times (fasting on the first day - at 07:45 a.m.; after the exercise session on the first day - at 11:00 a.m.; two hours postprandial on the first day - at 02:30 p.m.; fasting on the second day - at 08:30 a.m.) while participants spend 32 hours inside the whole body calorimetry unit while receiving a high-protein diet or a control diet.
Changes in blood insulin levels. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  Changes in insulin will be assessed four times (fasting on the first day - at 07:45 a.m.; after the exercise session on the first day - at 11:00 a.m.; two hours postprandial on the first day - at 02:30 p.m.; fasting on the second day - at 08:30 a.m.) while participants spend 32 hours inside the whole body calorimetry unit while receiving a high-protein diet or a control diet.
Changes in blood lipid panel levels. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  Changes in lipid panel will be assessed four times (fasting on the first day - at 07:45 a.m.; after the exercise session on the first day - at 11:00 a.m.; two hours postprandial on the first day - at 02:30 p.m.; fasting on the second day - at 08:30 a.m.) while participants spend 32 hours inside the whole body calorimetry unit while receiving a high-protein diet or a control diet.
Changes in blood peptide tyrosine-tyrosine levels. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  Changes in peptide tyrosine-tyrosine will be assessed four times (fasting on the first day - at 07:45 a.m.; after the exercise session on the first day - at 11:00 a.m.; two hours postprandial on the first day - at 02:30 p.m.; fasting on the second day - at 08:30 a.m.) while participants spend 32 hours inside the whole body calorimetry unit while receiving a high-protein diet or a control diet.
Changes in blood glucagon-like peptide-1 levels. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  Changes in glucagon-like peptide-1 will be assessed four times (fasting on the first day - at 07:45 a.m.; after the exercise session on the first day - at 11:00 a.m.; two hours postprandial on the first day - at 02:30 p.m.; fasting on the second day - at 08:30 a.m.) while participants spend 32 hours inside the whole body calorimetry unit while receiving a high-protein diet or a control diet.
Changes in blood ghrelin levels. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  Changes in ghrelin will be assessed four times (fasting on the first day - at 07:45 a.m.; after the exercise session on the first day - at 11:00 a.m.; two hours postprandial on the first day - at 02:30 p.m.; fasting on the second day - at 08:30 a.m.) while participants spend 32 hours inside the whole body calorimetry unit while receiving a high-protein diet or a control diet.
Changes in blood leptin levels. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  Changes in leptin will be assessed four times (fasting on the first day - at 07:45 a.m.; after the exercise session on the first day - at 11:00 a.m.; two hours postprandial on the first day - at 02:30 p.m.; fasting on the second day - at 08:30 a.m.) while participants spend 32 hours inside the whole body calorimetry unit while receiving a high-protein diet or a control diet.
Changes in blood free glycerol levels. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  Changes in glycerol will be assessed four times (fasting on the first day - at 07:45 a.m.; after the exercise session on the first day - at 11:00 a.m.; two hours postprandial on the first day - at 02:30 p.m.; fasting on the second day - at 08:30 a.m.) while participants spend 32 hours inside the whole body calorimetry unit while receiving a high-protein diet or a control diet.
Changes in blood free fatty acids levels. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  Changes in free fatty acids will be assessed four times (fasting on the first day - at 07:45 a.m.; after the exercise session on the first day - at 11:00 a.m.; two hours postprandial on the first day - at 02:30 p.m.; fasting on the second day - at 08:30 a.m.) while participants spend 32 hours inside the whole body calorimetry unit while receiving a high-protein diet or a control diet.
Difference in energy expenditure assessed by indirect calorimetry during 32 hours of a high-protein (HP) total diet replacement compared to 32hours of a control (CON) diet. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  To measure the differences in selected components of energy expenditure (resting, basal, sleep and postprandial - kcal) during 32 hours of a high-protein (HP) total diet replacement compared to 32 hours of a control (CON) diet.
Difference in substrate oxidation assessed by indirect calorimetry during 32 hours of a high-protein (HP) total diet replacement compared to 32hours of a control (CON) diet. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  To measure the differences in substrate oxidation rates (carbohydrate and protein - grams per day) during 32 hours of a high-protein (HP) total diet replacement compared to 32 hours of a control (CON) diet.
Difference in substrate balance assessed by indirect calorimetry during 32 hours of a high-protein (HP) total diet replacement compared to 32hours of a control (CON) diet. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  To measure the differences in substrate balance (carbohydrate and protein - grams per day) during 32 hours of a high-protein (HP) total diet replacement compared to 32 hours of a control (CON) diet.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Prado, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oliveira CLP, Boule NG, Elliott SA, Sharma AM, Siervo M, Berg A, Ghosh S, Prado CM. A high-protein total diet replacement alters the regulation of food intake and energy homeostasis in healthy, normal-weight adults. Eur J Nutr. 2022 Jun;61(4):1849-1861. doi: 10.1007/s00394-021-02747-1. Epub 2021 Dec 20. PMID 34928408
- [Derived] Oliveira CLP, Boule NG, Sharma AM, Elliott SA, Siervo M, Ghosh S, Berg A, Prado CM. A high-protein total diet replacement increases energy expenditure and leads to negative fat balance in healthy, normal-weight adults. Am J Clin Nutr. 2021 Feb 2;113(2):476-487. doi: 10.1093/ajcn/nqaa283. PMID 33247306
- [Derived] Oliveira CLP, Boule NG, Sharma AM, Elliott S, Siervo M, Ghosh S, Berg A, Prado CM. Examining the effects of a high-protein total diet replacement on energy metabolism, metabolic blood markers, and appetite sensations in healthy adults: protocol for two complementary, randomized, controlled, crossover trials. Trials. 2019 Dec 27;20(1):787. doi: 10.1186/s13063-019-3950-y. PMID 31881910